CLINICAL TRIAL: NCT06722950
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase II Clinical Study of AC591 in Preventing Oxaliplatin-Induced Peripheral Neuropathy
Brief Title: Phase II Clinical Study of AC591 in Preventing Oxaliplatin-Induced Peripheral Neuropathy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NTP-AC591-001; Shandong New Time Pharmaceutic (Other: Shandong New Time Pharmaceutical Co., Ltd.)
Record Dates: First submitted 2024-10-22; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Colorectal Adenoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AC591+CAPEOX (Experimental): AC591 granules (3 times a day) + CAPEOX chemotherapy
  Interventions: Drug: CAPEOX; Drug: AC591
- Placebo+CAPEOX (Placebo Comparator): Placebo (3 times a day) + CAPEOX chemotherapy
  Interventions: Drug: CAPEOX; Drug: Placebo

INTERVENTIONS:
Drug: CAPEOX — CAPEOX: 130mg/m2 of oxaliplatin (D1, central intravenous drip for 2h (time window + 20min)), 1000mg/m2 of capecitabine tablets each time, orally, twice a day (D1-D14, morning and evening); repeat the CAPEOX chemotherapy regimen every 3 weeks.
Drug: Placebo — Placebo：3 times a day (daily), taken with boiled water.
  Arms: Placebo+CAPEOX
Drug: AC591 — AC591 : 3 times a day (daily), taken with boiled water.
  Arms: AC591+CAPEOX

SUMMARY:
A randomized, double-blind, placebo-controlled, multicenter, Phase II clinical study of AC591 in preventing Oxaliplatin-Induced Peripheral Neuropathy

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind, placebo-controlled trial aims to explore the effectiveness of AC591 particles in preventing oxaliplatin-induced peripheral neuropathy. Patients with colorectal adenocarcinoma who are prepared to receive CAPEOX (capecitabine tablets + oxaliplatin injection) postoperative adjuvant chemotherapy within 3 weeks to 2 months after surgery will be randomized in a 1:1 ratio. The subjects will be stratified based on the chemotherapy cycles they are prepared to receive CAPEOX (4 cycles vs 8 cycles).

ELIGIBILITY:
Inclusion Criteria:

1. Understand the experimental procedures and contents, and voluntarily sign a written informed consent;
2. Male or female subjects aged 18 to 75 years (inclusive) when signing the informed consent;
3. Patients with histologically confirmed colorectal adenocarcinoma. Prepare to receive CAPEOX postoperative adjuvant chemotherapy within 3 weeks to 2 months after surgery, and have never used oxaliplatin;
4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1 before the first medication in the study;
5. Organ function level before the first medication in the study meets the following requirements:

   Peripheral blood cell count: white blood cell count ≥3×109/L and neutrophil ≥1.5×109/L, platelet count ≥75×109/L, hemoglobin ≥90g/L; Liver function: total bilirubin ≤1.5 times the upper limit of normal reference value; alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal reference value; Renal function: serum creatinine ≤1.5 times the upper limit of normal reference value.
6. Male or female subjects of fertility are required to take effective medical contraceptive measures until 3 months after the last study administration.

Exclusion Criteria:

1. known neurodegenerative disease (e.g., Parkinson's disease, Alzheimer's disease, Huntington's disease) or neuromuscular disease (e.g., multiple sclerosis, amyotrophic lateral sclerosis, poliomyelitis, hereditary neuromuscular disease);
2. Patients diagnosed with damp-heat syndrome or liver depression-fire syndrome according to TCM during the screening period;
3. Patients with severe diabetic peripheral neuropathy (such as muscle atrophy as the main stage) and abnormal electromyography;
4. Patients with known allergic reactions to any component of the study drug;
5. Patients with intestinal obstruction that requires treatment;
6. Active severe clinical infection (> grade 2, National Cancer Institute-Common Adverse Event Evaluation Criteria [NCI-CTCAE V5.0]), including active tuberculosis;
7. Uncontrolled diabetes, severe lung disease (such as acute lung disease, pulmonary fibrosis affecting lung function, interstitial lung disease, but excluding recovered radiation pneumonia), liver failure;
8. Clinically significant cardiovascular disease, New York Heart Association [NYHA] grade III-IV congestive heart failure, unstable angina, myocardial infarction, etc. within 6 months before the first dose. Uncontrolled hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg after adequate treatment);
9. Patients who need to take coumarin derivative anticoagulants (such as warfarin, phenprocoumon) regularly within 3 weeks before screening or during the study;
10. Patients who have used drugs that interfere with the evaluation of neuropathic pain (such as antidepressants, antiepileptic drugs) within 2 weeks before the first dose;
11. Renal replacement therapy;
12. Previous history of organ transplantation, autologous/allogeneic stem cell transplantation;
13. History of other malignant tumors except colorectal cancer in the past 5 years. However, cured basal cell carcinoma of the skin, carcinoma in situ of the cervix, or early papillary thyroid carcinoma are excluded;
14. HIV infection, hepatitis B surface antigen positive (and peripheral blood hepatitis B virus deoxynucleotide HBV DNA ≥ 1×104 copies/mL or ≥ 2000IU/mL), hepatitis C virus antibody positive (and peripheral blood hepatitis C virus nucleotide HCV RNA ≥ 1×103 copies/ml or ≥ 200IU/mL) or active syphilis patients;
15. Pregnancy (confirmed by menstrual pregnancy test) or lactation;
16. Current alcohol or drug dependence;
17. Suffering from known mental illness disorders that may affect trial compliance;
18. Adverse events of previous anti-tumor treatment have not recovered to grade 1 (NCI-CTCAE V5.0) or abnormalities have no clinical significance;
19. Subjects who have participated in other interventional clinical trials within 4 weeks before the first study drug;
20. The investigator believes that the patient has other factors that affect the efficacy or safety evaluation of this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with grade 1-3 oxaliplatin-induced peripheral neuropathy as assessed by the oxaliplatin-specific Levi rating tool | At the end of Cycle 4 （each cycle is 21 days）

SECONDARY OUTCOMES:
Proportion of subjects with grade 1-3 oxaliplatin-induced peripheral neuropathy as assessed by the oxaliplatin-specific Levi rating tool | At the end of Cycle 8（each cycle is 21 days）
The time of onset of grade 1-3 oxaliplatin-induced peripheral neuropathy assessed by the Levi rating tool for oxaliplatin | At the end of Cycle 4 and 8（each cycle is 21 days）
The incidence of NCI-CTCAE V5.0 ≥ grade 2 neurotoxicity in subjects during CAPEOX chemotherapy | At the end of Cycle 4 and 8（each cycle is 21 days）
The change in the EORTC-QLQ-CIPN20 score of subjects during CAPEOX chemotherapy from baseline | at the end of each cycle（each cycle is 21 days）
The change in the EORTCQLQ-C30 score of subjects during CAPEOX chemotherapy from baseline | At the end of Cycle 4 and 8（each cycle is 21 days）
The proportion of subjects who used analgesics due to peripheral neuropathy caused by CAPEOX chemotherapy | At the end of Cycle 4 and 8（each cycle is 21 days）
The proportion of subjects who developed acute peripheral neuropathy within 3 days after the first CAPEOX chemotherapy | At the end of Cycle 4 and 8（each cycle is 21 days）
The average cumulative dose of oxaliplatin received by the subjects during CAPEOX chemotherapy | At the end of Cycle 4 and 8（each cycle is 21 days）
The incidence of gastrointestinal adverse reactions in the subjects during CAPEOX chemotherapy | At the end of Cycle 4 and 8（each cycle is 21 days）
The proportion of subjects who did not experience neurotoxicity as assessed by the Levi rating tool dedicated to oxaliplatin | At the end of Cycle 4 and 8（each cycle is 21 days）

IPD SHARING:
Plan to Share IPD: No